CLINICAL TRIAL: NCT02974842
Title: Cytological Evaluation of Specimens Collected With the MAKO 7 Device in Pre Salpingo-Oophorectomy Subjects for Determination and/or Differentiation of Normal Versus Atypical Versus Malignant Cells
Brief Title: Pre-Salpingo-Oophorectomy Pilot Study of MAKO 7 Device Performance
Status: Completed | Type: Observational
Sponsor: nVision Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN 0276
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; Atypia Suspicious for Malignancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cell samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-Salpingo-Oophorectomy: Women with pelvic mass suspicious for malignancy or have BRCA1 or BRCA2 mutations that will undergo pre-salpingo-oophorectomy.
  Interventions: Device: MAKO 7

INTERVENTIONS:
Device: MAKO 7 — Hysteroscopic cell sampling

SUMMARY:
This study evaluates the ability of the MAKO 7 device to collect various cells

DETAILED DESCRIPTION:
Prospective, multi-center observational study to evaluate the ability of the MAKO 7 device to collect cells from the fallopian tubes for cytological evaluation for determination and/or differentiation of normal versus atypical versus malignant cells.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is medically cleared for surgery
2. Subject is scheduled to undergo a salpingo-oophorectomy for a pelvic mass suspicious for malignancy or for BRCA1 or BRCA2 mutations
3. Subject must be 18 years of age
4. Subject must be able to provide informed consent

Exclusion Criteria:

1. Contraindication to hysteroscopy
2. Acute pelvic inflammatory disease
3. Active or recent lower pelvic infection
4. Pregnancy
5. Delivery or termination of a pregnancy in the past 6 weeks
6. Known tubal obstruction including tubal ligation
7. Invasive carcinoma of the cervix or endometrium
8. Intolerance of anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with pelvic mass suspicious for malignancy or have BRCA1 or BRCA2 mutations that put them at high risk of developing malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Sarna, B.S., Study Director — nVision Medical Corp
Locations (3):
- United States (3):
  - Kaiser Permanente, San Francisco, California
  - Kaiser Permanente, Walnut Creek, California
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women scheduled for a salpingo-oophorectomy surgery due to suspicious adnexal mass or due to BRCA 1 or BRCA 2 mutation were recruited from three gynecologic oncology centers in the United States.
Pre-assignment Details: This was a single arm study evaluating the feasibility of a novel hysteroscopic catheter to collect cytological samples.
Groups:
- MAKO 7 Group: Women scheduled for a salpingo-oophorectomy surgery due to suspicious adnexal mass or due to BRCA 1 or BRCA 2 mutation.
Period: Overall Study
Arm/Group | MAKO 7 Group
Started | 50 (Participants)
Completed | 42
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Screen failures | 4

BASELINE CHARACTERISTICS:
Groups:
- Eligible Participants With Hysteroscopic Attempt: Women scheduled for salpingo-oophorectomy who provided consent and met all inclusion criteria and none of the exclusion criteria.
Arm/Group | Eligible Participants With Hysteroscopic Attempt
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 6
  Race/Ethnicity: Caucasian | 29
  Race/Ethnicity: Hispanic or Latino | 3
  Race/Ethnicity: Native American or other Pacific Islander | 1
  Race/Ethnicity: Non-Hispanic or non-Latino | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Reason for Surgery [Count of Participants; unit: Participants]
  Pelvic mass suspicious for malignancy | 34
  BRCA 1 or BRCA 2 mutations | 8

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Cytological Findings From Fallopian Tubes to Surgical Histology Results.
Description: Cytological evaluations of samples collected from fallopian tubes were performed in a blinded fashion to histology findings from excised fallopian tubes and ovaries. Concordance was evaluated between cytology where collected samples were adequate and available histology.
Time Frame: Up to 60 days post-operatively
Population: Fallopian tubes with adequate samples for cytological evaluation and available surgical histology results.
Measure: Count of Units; unit: fallopian tubes
Units Other Than Participants: fallopian tubes
Groups:
- MAKO 7 Group: Fallopian tubes with adequate cytology samples obtained with MAKO 7 with available surgical histology results.
Arm/Group | MAKO 7 Group
Number analyzed (Participants) | 29
Number analyzed (fallopian tubes) | 44
fallopian tubes
  Concordant | 42
  Discordant | 2

ADVERSE EVENTS:
Time Frame: Study procedure or device related adverse events were recorded until 24 hours post study procedure or until discharge, whichever happened first.
Groups:
- MAKO 7 Group: Women scheduled for salpingo-oophorectomy who provided consent and met all inclusion criteria.
Arm/Group | MAKO 7 Group
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 25/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAKO 7 Group (N=42)
Uterine perforation (Reproductive system and breast disorders) | 3 (3)
Nausea (General disorders) | 7 (8) — Not related to study procedure or study device
Pain (Surgical and medical procedures) | 22 (24) — Not related to study procedure or study device
Dizziness (General disorders) | 4 (4) — Not related to study procedure or study device
Fatigue (General disorders) | 7 (7) — Not related to study procedure or study device
Hypotension (General disorders) | 6 (7) — Not related to study procedure or study device
Anemia (Blood and lymphatic system disorders) | 11 (11) — Not related to study procedure or study device
Hematological Dyscrasia (Blood and lymphatic system disorders) | 7 (10) — Not related to study procedure or study device
Electrolyte Imbalance (General disorders) | 7 (9) — Not related to study procedure or study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02974842/Prot_SAP_000.pdf